CLINICAL TRIAL: NCT00430352
Title: A Study to Evaluate the Safety of MabThera (Rituximab) Maintenance Therapy in Patients With Follicular Non-Hodgkin's Lymphoma Who Have Responded to Induction Therapy.
Brief Title: MAXIMA Study: A Study of Maintenance Therapy With MabThera (Rituximab) in Patients With Non-Hodgkin's Lymphoma.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO19872
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 375mg/m2 iv every 8 weeks

SUMMARY:
This single arm study will evaluate the safety and efficacy of MabThera maintenance therapy following a MabThera-containing induction regimen in first line or relapsed patients with follicular non-Hodgkin's lymphoma. All patients will receive MabThera 375mg/m2 body surface area, as an intravenous infusion, every 8 weeks. The anticipated time on study treatment is 1-2 years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically confirmed grade 1, 2 or 3a follicular non-Hodgkin's lymphoma;
* patients who have received adequate (>=8 cycles) induction therapy with MabThera as first line treatment, or treatment for relapsed disease;
* demonstrated partial or complete response to induction therapy.

Exclusion Criteria:

* stable or progressive disease after most recent induction therapy;
* transformation to high grade lymphoma;
* patients with prior or concomitant malignancies, except non-melanoma skin cancer or adequately treated in situ cancer of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2006-09-04 (Actual); Primary Completion 2011-05-26 (Actual); Study Completion 2011-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (178):
- University "Mother Theresa" Hospital Center; Oncology Department, Tirana, Albania
- Argentina (8):
  - Instituo Lavalle de Oncologia; Hematology, Bahía Blanca
  - Academia Nacional de Medicina; Inst. de Cardiologia, Buenos Aires
  - Fundaleu; Haematology, Buenos Aires
  - Hospital Churruca Visca; Haematology, Buenos Aires
  - Hospital Jr Vidal; Jefe de Servicio de Clinica Medica/Hematologia, Corrientes
  - Sanatorio Allende; Haematology, Córdoba
  - HOSPITAL PRIVADO - CENTRO MEDICO DE CÓRDOBA; Dpto Oncología, Córdoba
  - Hospital General San Martin; Haematology, La Plata
- Australia (5):
  - Liverpool Hospital; Haematology, Liverpool, New South Wales
  - Wollongong Hospital; Cancer Services, Wollongong, New South Wales
  - Royal Brisbane Hospital; Oncology Department, Brisbane, Queensland
  - Haematology & Oncology Clinics of Australia, Mater Medical Centre, South Brisbane, Queensland
  - Mount Medical Center, Perth, Western Australia
- Bosnia and Herzegovina (4):
  - University Clinical Center of the Republic of Srpska, Clinic for Internal Disease, Hematology Dept, Banja Luka
  - Inst. of Hematology, Kasindo
  - Uni Hospital Mostar, Mostar
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (13):
  - CEHON, Salvador, Estado de Bahia
  - Nucleo de Oncologia da Bahia - NOB, Salvador, Bahia, Estado de Bahia
  - ONCOMED, Belo Horizonte, Minas Gerais
  - Centro de Tratamento Oncologico - Oncoclinica, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UFRGS; Medicina Interna, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Hospital das Clinicas - UNICAMP; Hemoterapia, Campinas, São Paulo
  - Clinica Oncologica De Piracicaba Sc, Piracicaba, São Paulo
  - Hospital Alemao Oswaldo Cruz; Oncologia, São Paulo, São Paulo
  - Hospital Estadual do Servidor Publico; Hematologia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP, Oncologia, São Paulo, São Paulo
- Bulgaria (5):
  - UMHAT Dr Georgi Stranski; Hematology, Pleven
  - Umhat S. George; Hematology, Plovdiv
  - UMHAT Alexandrovska EAD; Hematology, Sofia
  - National Center of Hematology & Transfusiology; Clinical Unit, Clinic of Hematology, Sofia
  - Mhat Sveta Marina; Dept. of Haematology, Varna
- Colombia (2):
  - Centro Médico Carlos Ardila Lule, Bucaramanga
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
- Croatia (3):
  - Clinical Hospital Centre Split; Dept Of Hematology, Split
  - Clinical Hospital Centre Dubrava; Hematology Department, Zagreb
  - University Hospital Center Zagreb; Haematology Department, Zagreb
- Ecuador (2):
  - Hospital José Carrasco; Oncology Service, Cuenca
  - Hospital Carlos Andrade Marin; Servicio de Oncología, Quito
- Oncology & Radiotherapy Centre; Oncology, Cairo, Egypt
- Finland (4):
  - Kanta-Hämeen Keskussairaala; Dept of Internal Medicine, Hematology, Hämeenlinna
  - Kymenlaakson keskussairaala, Kotka
  - Päijät-Hämeen Keskussairaala; Dept of Internal Medicine, Hematology, Lahti
  - Satakunnan Keskussairaala; Sisaetauti Osasto, Pori
- Germany (25):
  - Internist; Praxis Für Haemotologie & Onkologie, Bad Soden
  - Dres.Christian Sperling und Claudia Schelenz, Berlin
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Universitätsklinikum Bonn; Medizinische Klinik und Poliklinik I; Allgemeine Innere Medizin, Bonn
  - Dres. Matthias Adler Oliver Marschal und Andreas Pies, Braunschweig
  - Gemeinschaftspraxis, Duisburg
  - Internistische Praxis Dr. Plingen, Düsseldorf
  - Internistische Schwerpunktpraxis Erlangen, Erlangen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Onkologische Gemeinschaftspraxis, Prof. Dr. Gropp, Dr. Depenbusch und Dr. Rösel, Gütersloh
  - Überörtliche Gemeinschaftspraxis Schwerpunkt Hämatologie, internistische Onkologie & Palliativmed., Hamburg
  - Onkologische Schwerpunktpraxis; Herrn Dr. Med. Bertram, Hamburg
  - Dres.Andreas Karcher und Stefan Fuxius, Heidelberg
  - Uniklinik Heidelberg, Medizinische Klinik & Poliklinik V, Heidelberg
  - Onkologische Schwerpunktpraxis (Eps-Gmbh), Jena
  - Märkische Kliniken GmbH, Klinikum Lüdenscheid; Hämatologie / Onkologie, Lüdenscheid
  - Stauferklinikum Schwäb.Gmünd, Mutlangen
  - Gemeinschaftspraxis Dres. Schröder, Sieg, Mülheim
  - Onko. Gemeinschaftspraxis Dres. Tigges/ Böning/ Abenhardt/ Bosse, München
  - Dres.Ulrich Hutzschenreuter und Uwe Sauer, Nordhorn
  - Onkologische Praxis Oldenburg; Dres. Otremba, Reschke, Zirpel, Kühn und Ruff, Oldenburg
  - Praxis für Onkologie und Hämatologie, Recklinghausen
  - Diakonie-Klinikum Klinik für Innere Medizin III Abt.Hämatologie, intern. Onkologie und Palliativmedi, Schwäbisch Hall
  - Internistische Gemeinschaftspraxis Dres. Hoering/Von Ehr/Responde, Stuttgart
  - Haematologisch-Onkologische Praxis; Dr. med. Christoph Maintz und Matthias Groschek, Würselen
- Greece (3):
  - Laiko General Hospital - Uni of Athens; 1St Dept. of Internal Medicine, Athens
  - Attiko Hospital; Haematology Clinic, Athens
  - Theagenio Anticancer Hospital; Dept. of Haematology, Thessaloniki
- Israel (5):
  - Rambam Medical Center; Heamatology & Bone Marrow Transplantation, Haifa
  - Wolfson Mc; Haematology, Holon
  - Hadassah Ein Karem Hospital; Haematology, Jerusalem
  - Chaim Sheba Medical Center; Hematology BMT & CBB, Ramat Gan
  - Ichilov Sourasky Medical Center; Heamatology, Tel Aviv
- Italy (39):
  - Ospedale Civile Dello Spirito Santo; Divisione Di Ematologia, Pescara, Abruzzo
  - Uni Degli Studi Di Bari, Policlinico; Cattedra Di Ematologia,Dipart. Di Medicina Interna E Publica, Bari, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - Az. Osp. C. Panico; Rep. Ematologia E Trapianto, Tricase - Le, Apulia
  - Az. Osp. Pugliese; Dh Oncologico, Catanzaro, Calabria
  - Ospedale S. Gennaro; Divisione Di Ematologia, Napoli, Campania
  - Ospedale Cardarelli; Divisione Di Ematologia, Napoli, Campania
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - Arcispedale S. Anna; Sezione Di Ematologia, Ferrara, Emilia-Romagna
  - A.O. Universitaria Policlinico Di Modena; Ematologia, Modena, Emilia-Romagna
  - A.O.U. Policlinico di Modena-Dipartimento di Medicina Diagnostica, Clinica e di Sanità pubblica, Modena, Emilia-Romagna
  - Irccs Centro Di Riferimento Oncologico (CRO); Dipartimento Di Oncologia Medica, Aviano, Friuli Venezia Giulia
  - Az. Osp. Uni Ria Policlinico Tor Vergata; Unita Di Ematologia, Rome, Lazio
  - Ospedale S. Eugenio; Divisione Di Ematologia, Rome, Lazio
  - Univ. Cattolica La Sapienza; Cattedra Di Ematologia, Rome, Lazio
  - Uni Cattolica; Divisione Di Ematologia, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova; Ematologia 1, Genoa, Liguria
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili;U.O. Ematologia, Brescia, Lombardy
  - Istituto S. Raffaele Monte Tabor; Divisione Ematologia E Utmo, Milan, Lombardy
  - Ist. Nazionale Per Lo Studio E Cura Dei Tumori; Div. Ematologia Trapianto Midollo Osseo Allogenico, Milan, Lombardy
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - ASST DI MONZA; Ematologia, Monza, Lombardy
  - Irccs Policlinico San Matteo; Divisione Di Ematologia, Pavia, Lombardy
  - Fondazione Del Piemonte Per L'oncologia Ircc Di Candiolo; Dipartimento Oncologico, Candiolo, Piedmont
  - Az. Osp. S. Croce Ospedale Generale; Sezione Di Ematologia, Cuneo, Piedmont
  - Univ. Piemonte Est Amedeo Avogadro; Div.Ematologia- Dip.Clinica Med.Sperim.& Ircad, Novara, Piedmont
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino; Ematologia 1, Turin, Piedmont
  - A.O.U. Citta' Della Salute E Della Scienza-P.O. Molinette;S.C. Ematologia, Turin, Piedmont
  - Ospedale Oncologico A Businco-Cagliari; Ematologia Sez., Cagliari, Sardinia
  - Ospedale V. Cervello; U.O. Ematologia E Trapianti, Palermo, Sicily
  - Ospedale Ferrarotto; Divisione Di Ematologia, Via S. Sofia 78, Sicily
  - Ospedale Civile; S.C. Ematologia, Pesaro, The Marches
  - A.O. Univ.Ospedali Riuniti Umerto I -G.M.Lancisi G.Salesi; U.O. Clinica Di Ematologia, Torrette Di Ancona, The Marches
  - Az. Osp. Di Careggi; Divisione Di Ematologia, Florence, Tuscany
  - Ospedale Santa Chiara; Unita Operativa Di Ematologia, Pisa, Tuscany
  - A.O. Universitaria Senese; Ematologia, Siena, Tuscany
  - Azienda Ospedaliera S. Maria della Misericordia; Ematologia, Perugia, Umbria
  - Uni Degli Studi; Dip.Med.Clinica E Sperim. Ematologia, Padua, Veneto
  - Ospedale Di Vicenza; Nefrologia, Ematologia, Vicenza, Veneto
- Mexico (7):
  - Issste; Haematology, Chihuahua City
  - Hospital Cima (Centro Internacional de Medicina) ; Haematology, Chihuahua City
  - Hospital Central de Pemex Norte Azcapotzalco, Mexico City
  - Hospital Español de Mexico, Mexico City
  - Hospital Regional Issste; Oncologia, Monterrey
  - Clinca San Jose; Haematology, Obregón
  - Issstep Puebla, ; Haematology, Puebla City
- Romania (6):
  - Spitalul Clinic Judetean de Urgenta Brasov,Clinica de Hematologie, Brasov
  - Fundeni Clinical Inst. ; Hematology Dept, Bucharest
  - Spitalul Clinic Coltea; Clinica de Hematologie, Bucharest
  - Oncology Inst. Cluj-Napoca; Cancer Dept, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sf. Spiridon Iasi, Clinica de Hematologie, Iași
  - Spitalul Clinic Judetean de Urgenta Targu-Mures; compartiment Hematologie, Târgu Mureş
- Russia (16):
  - Regional Clinical Hospital; Hematology, Belgorod
  - Clinical Oncology Dispensary of Ministry of Health of Tatarstan, Kazan'
  - Blokhin Cancer Research Center; Clinical Oncology, Moscow
  - City Clinical Hospital After Botkin; Hematology, Moscow
  - Vladimirskiy Regional Scientific Research Inst. ; Hematology, Moscow
  - Regional Clinical Hospital N.A. Semashko; Hematology, Nizhny Novgorod
  - City Hematological Center of Clinical Hospital #2; Hematology, Novosibirsk
  - Rostov State Medical Uni ; Hematology, Rostov-on-Don
  - Research Inst. of Hematology & Blood Transfusion ; Hematology, Saint Petersburg
  - Pavlov State Medical Uni ; Bone Marrow Transplantation Clinic, Saint Petersburg
  - Leningrad Regional Clinical Hospital; Hematology #1, Saint Petersburg
  - Stavropol Clinical Oncology Dispansary, Stavropol
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa
  - Ulyanovsk Regional Oncology Dispensary; Chemotherapy, Ulyanovsk
  - Regional Oncology Center; Chemotherapy, Volgograd
  - Regional Clinical Hospital; Hematology, Yaroslavl
- Slovakia (4):
  - Fakultna Nemocnica Roosevelta; Dept. of Haematology, Banská Bystrica
  - National Oncology Inst. ; Dept. of Haematology, Bratislava
  - Uni Hospital; Clinic of Haematology, Košice
  - Uni Hospital ; Dept. of Haematol. & Transfusion Medicine, Martin
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- Spain (9):
  - Hospital General de Castellon; Servicio de Hematologia, Castellon, Castellon
  - Complejo Asistencial Universitario De Burgos; Servicio de Oncologia, Burgos
  - Hospital Generla de Ciudad Real; Servicio de Oncologia, Ciudad Real
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Hospital El Bierzo; Servicio de Oncologia, León
  - Hospital Costa del Sol; Servicio de Hematologia, Málaga
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen Macarena; Servicio de Hematologia, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
- Sweden (6):
  - Laenssjukhuset; Medicinkliniken/Hematologsektionen, Halmstad
  - Sunderby Sjukhus; Medicinkliniken, Luleå
  - Skånes Universitetssjukhus; Kliniska Forskningsenheten Onkologimottagning medicinsk behandling, Malmo
  - Länssjukhuset Sundsvall-Härnösand, Medicinkliniken, Sundsvall
  - Uddevalla Sjukhus; Medicinkliniken, Uddevalla
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Switzerland (4):
  - Andreas Klinik; Onko-Hämatologisches Zentrum Cham Zug, Cham
  - Kantonsspital Graubünden;Onkologie und Hämatologie, Chur
  - Clinica Santa Chiara; Oncologia / Ematologia, Locarno
  - UniversitätsSpital Zürich; Zentrum für Hämatologie und Onkologie, Klinik für Onkologie, Zurich
- Turkey (Türkiye) (5):
  - Ankara Numune Egitim Ve Arastirma Hastanesi; Hematoloji Klinigi, Ankara
  - Hacettepe Uni Medical Faculty; Hematology, Ankara
  - Gazi Uni Medical School; Hematology, Ankara
  - Istanbul Uni Capa Hospital; Hematology, Istanbul
  - Ege Uni Medical School; Hematology, Izmir

REFERENCES:
- [Derived] Witzens-Harig M, Foa R, Di Rocco A, van Hazel G, Chamone DF, Rowe JM, Arcaini L, Poddubnaya I, Ho AD, Ivanova V, Vranovsky A, Thurley D, Oertel S. Maintenance with rituximab is safe and not associated with severe or uncommon infections in patients with follicular lymphoma: results from the phase IIIb MAXIMA study. Ann Hematol. 2014 Oct;93(10):1717-24. doi: 10.1007/s00277-014-2103-3. Epub 2014 May 14. PMID 24824768

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 375 Milligrams Per Square Meter (mg/m^2): Participants received rituximab 375 mg/m^2 intravenously (IV) once every 8 weeks for a total 12 infusions until progression, relapse, start of a new treatment, death, or toxicity.
Period: Overall Study
Arm/Group | Rituximab 375 Milligrams Per Square Meter (mg/m^2)
Started | 545
Completed | 407
Not Completed | 138
Not completed — Disease progression | 58
Not completed — Withdrawal by Subject | 11
Not completed — Adverse Event | 16
Not completed — Death | 5
Not completed — Other | 48

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all participants who completed a baseline visit and at least 1 further assessment.
Groups:
- Rituximab 375 mg/m^2: Participants received rituximab 375 mg/m^2 IV for up to 12 infusions in total every 8 weeks until progression, relapse, start of a new treatment, death, or toxicity.
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 313
  Male | 232

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE) - Overall Summary
Description: Data presented include percentage of participants with any AE, any infusion-related AE, any serious adverse event (SAE), any infusion-related SAE (counted separately from SAEs), death, and participants with toxicity as the primary cause for treatment discontinuation.
Time Frame: 24 months
Population: Safety Population: any participant who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 534
percentage of participants
  Any AE | 67.4
  Any infusion-related AE | 5.8
  Any non-infusion related SAE | 20.2
  Any infusion-related SAE | 0.2
  Deaths | 7.5
  Toxicity as primary cause for discontinuation | 3.0

2. Secondary Outcome: Progression-Free Survival - Percentage of Participants With an Event
Description: PFS was measured from the day of first rituximab maintenance infusion until the date of first documented disease progression or death by any cause. Participants who experienced none of these events at the time of analysis (clinical cutoff) and participants who were lost to follow-up were censored at their last clinical assessment date.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants | 24.0

3. Secondary Outcome: Progression-Free Survival - Time to Event
Description: as for outcome 2
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
months | NA [NA to NA] — Median and 95 percent (%) confidence interval (CI) for PFS could not be estimated due to the large number of censored participants and the short duration of follow-up.

4. Secondary Outcome: Event-Free Survival (EFS) - Percentage of Participants With an Event
Description: The percentage of participants who experienced PD or death or required a next or new lymphoma treatment over a study period of 2 years with 1 year of follow-up. EFS was measured from the day of first rituximab maintenance infusion until the date of first documented disease progression, death by any cause, or the institution of new anti-lymphoma treatment. Participants who experienced none of these events at the end of the study and participants who were lost to follow-up were censored at their last clinical assessment date.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants | 24.4

5. Secondary Outcome: Event-Free Survival (EFS) - Time to Event
Description: EFS was measured from the day of first rituximab maintenance infusion until the date of first documented disease progression, death by any cause, or the institution of new anti-lymphoma treatment. Participants who experienced none of these events at the end of the study and participants who were lost to follow-up were censored at their last clinical assessment date.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
months | NA [NA to NA] — Median and 95% CI for EFS could not be estimated due to the large number of censored participants and the short duration of follow-up.

6. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: As a measure of overall survival (OS), the percentage of participants who died over the study period of 2 years with 1 year of follow-up. OS was determined from the day of first rituximab maintenance infusion until the date of death irrespective of cause. Participants who had not died at the time of end of the whole study and participants who were lost to follow up were censored at the date of the last contact.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants | 7.3

7. Secondary Outcome: Overall Survival (OS) - Time to Event
Description: OS was determined from the day of first rituximab maintenance infusion until the date of death irrespective of cause. Participants who had not died at the time of end of the whole study and participants who were lost to follow up were censored at the date of the last contact.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants | NA [NA to NA] — Median and 95% CI for OS could not be estimated due to the large number of censored participants and the short duration of follow-up.

8. Secondary Outcome: Time to Next Lymphoma Treatment (NLT) - Percentage of Participants With an Event
Description: As a measure of time to NLT (TNLT), the percentage of participants with new lymphoma treatment over a study period of 2 years with 1 year of follow-up. TNLT was measured from the date of first rituximab maintenance infusion to the date of first documented intake of any new anti-lymphoma treatment (chemotherapy, radiotherapy, immunotherapy, etc). Participants who did not have documentation that an NLT had started and participants who were lost to follow up were censored at their last visit where the assessment for start of any new lymphoma medication was actually made.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants | 17.4

9. Secondary Outcome: Time to NLT - Time to Event
Description: TNLT was measured from the date of first rituximab maintenance infusion to the date of first documented intake of any new anti-lymphoma treatment (chemotherapy, radiotherapy, immunotherapy, etc). Participants who did not have documentation that an NLT had started and participants who were lost to follow up were censored at their last visit where the assessment for start of any new lymphoma medication was actually made.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
months | NA [NA to NA] — Median and 95% CI for time to NLT could not be estimated due to the large number of censored participants and the short duration of follow-up.

10. Secondary Outcome: Percentage of Participants With Response by Best Response to Study Treatment
Description: Percentage of participants with complete response (CR), unconfirmed CR (CRu), no change, or progressive disease (PD). For each participant, the last response to induction therapy immediately prior to study entry was compared to the best response observed during rituximab maintenance therapy. Where possible, assessment of response was based on the International Workshop to Standardize Response Criteria for Non-Hodgkin's Lymphoma (NHL).
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population; only participants who received any study treatment were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 545
percentage of participants
  CR/CRu | 2.1
  No change | 87.5
  PD | 10.5

11. Secondary Outcome: Percentage of Participants With PR Who Converted to CRu
Description: Percentage of participants with PR or CR(u) conversion while on rituximab maintenance therapy over a study period of 2 years with 1 year of follow-up. For each participant, the last response to induction therapy immediately prior to study entry was compared to the best response observed during rituximab maintenance therapy. Assessment and definition of response was based on the International Workshop to Standardize Response Criteria for NHL.
Time Frame: Baseline, every 8 weeks during treatment, and 3, 6, 9 and 12 months after last dose
Population: ITT population; only participants with PR to most recent treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 161
percentage of participants | 6.2 [3.0 to 11.1]

ADVERSE EVENTS:
Time Frame: AEs were collected at up through 12 months after last dose (1 year follow-up).
Description: AEs were collected at up through 12 months after last dose (1 year follow-up). AEs occuring within 24 hours of infusion were considered infusion-related reactions (IRRs) and were collected and reported as separate events mutually exclusive from all 'other' AEs collected and reported. These events appear in the table labeled as 'IRR'.
Arm/Group | Rituximab 375 mg/m^2
Serious Adverse Events (participants affected / at risk) | 109/534
Other Adverse Events (participants affected / at risk) | 207/534
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=534)
Cerebrovascular accident - IRR (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 7
Appendicitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 2
Abdominal abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Aspergilloma (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cerebral aspergillosis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Meningitis enteroviral (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Coeliac disease (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Coronary artery disease (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Left ventricular dysfunction (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Palpitation (Cardiac disorders) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Osteosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 3
Cerebral ischaemia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Thalamus haemorrhage (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Pyrexia (General disorders) | 4
Chest pain (General disorders) | 2
Fatigue (General disorders) | 1
Sudden death (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Female sterilisation (Surgical and medical procedures) | 1
Finger amputation (Surgical and medical procedures) | 1
Inguinal hernia repair (Surgical and medical procedures) | 1
Small intestinal resection (Surgical and medical procedures) | 1
Cataract (Eye disorders) | 1
Eye haemorrhage (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Vascular occlusion (Vascular disorders) | 1
Depressed mood (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pregnancy of partner (Social circumstances) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=534)
Nasopharyngitis (Infections and infestations) | 38
Diarrhoea (Gastrointestinal disorders) | 31
Back pain (Musculoskeletal and connective tissue disorders) | 35
Arthralgia (Musculoskeletal and connective tissue disorders) | 34
Fatigue (General disorders) | 40
Pyrexia (General disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 50
Headache (Nervous system disorders) | 31
Hypertension (Vascular disorders) | 32
Blood lactate dehydrogenase increased (Investigations) | 37
Neutrophil count decreased (Investigations) | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.